CLINICAL TRIAL: NCT01404598
Title: A Phase 1 Study to Assess the Pharmacokinetics of Nitrates and Gamma-Hydroxybutyric Acid (GHB) After Oral Administration of Therapeutic and Supratherapeutic Doses of Naproxcinod in Healthy Male Subjects
Brief Title: Pharmacokinetics Study: Determination of Naproxcinod and Its Metabolites After Oral Administration in Male
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: NicOx, NicOx
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HCT 3012-X-114
Record Dates: First submitted 2011-06-16; First posted 2011-07-28 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — naproxen-n-butyl nitrate; Naproxen; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- naproxcinod 750 mg bid (Experimental)
  Interventions: Drug: naproxcinod 750 bid
- naproxcinod 3000 mg od (Experimental)
  Interventions: Drug: naproxcinod 3000 mg od
- naproxen 500 mg bid (Active Comparator)
  Interventions: Drug: naproxen 500 mg bid

INTERVENTIONS:
Drug: naproxcinod 750 bid — naproxcinod 750 bid
  Arms: naproxcinod 750 mg bid
Drug: naproxcinod 3000 mg od — naproxcinod 3000 mg od
  Arms: naproxcinod 3000 mg od
Drug: naproxen 500 mg bid — naproxen 500 mg bid
  Arms: naproxen 500 mg bid

SUMMARY:
This study will be performed in 2 parts conducted in parallel:

Part 1 (conducted on 16 healthy subjects): Administration of naproxcinod 750 mg or naproxen 500 mg twice a day (bid) during 7 days The main aim of this study part will be to assess the pharmacokinetic profile (i.e. the absorption, the distribution, the metabolism and the elimination of the drug after its administration) of nitrates (metabolite of naproxcinod) present in plasma, saliva and urine after oral administration of naproxcinod 750 mg bid for 7 days or naproxen 500 mg bid for 7 days as a reference.

Part 2 (conducted on 8 healthy subjects): Administration of a single dose of naproxcinod 3000 mg. The main aim of this study part will be to assess the pharmacokinetic profile (i.e. the absorption, the distribution, the metabolism and the elimination of the drug after its administration) of Gamma-Hydroxybutyric Acid (GHB), a compound resulting from the transformation of the naproxcinod, after oral administration of a single supratherapeutic dose of 3000 mg.

ELIGIBILITY:
Inclusion Criteria:1.

1. Healthy, non smoker male subjects aged 18 to 45 years (inclusive).
2. Body Mass Index (BMI) between 18 and 30 kg/m² (inclusive) with body weight (BW) ≥ 50 kg.
3. Normal physical examination (non clinically significant abnormalities), as judged by the investigator.
4. Normal electrocardiogram (ECG) (12-lead), (non clinically significant abnormalities), as judged by the Investigator.
5. Supine Systolic Blood Pressure (SBP) between 100 and 139 mmHg (inclusive) and Diastolic Blood Pressure (DBP) between 50 and 89 mmHg (inclusive) (mean of 3 measurements).
6. Supine Heart Rate (HR) between 45 and 90 bpm (inclusive).
7. Oral body temperature (BT) between 36 and 37.5°C (inclusive).
8. Subject must be able to understand the written information sheet and informed consent and comply with all study requirements.
9. Subject must provide a written, dated and signed informed consent prior to any study procedure.

Exclusion Criteria:

1. History of hypersensitivity reactions (such as asthma, rhinitis, or urticaria) to aspirin, naproxen or any other non steroidal anti-inflammatory drugs (NSAIDs); or hypersensitivity or contraindications to organic nitrate drugs; or to L-proline.
2. History of any clinically relevant gastrointestinal (such as gastritis or gastric ulcer), respiratory, psychiatric, neurologic, kidney, liver, cardiac disease, bleeding disorder, other disease/condition or abnormal physical finding which may interfere with the study objectives, as judged by the Investigator.
3. After 1 minute in a standing position, a drop of more than 20 mmHg in SBP or 10 mmHg in DBP compared to supine position (mean of 3 measurements) and a clinical manifestation of postural hypotension.
4. Any clinically significant abnormal laboratory values, including creatinine clearance ≤ 80 mL/min as calculated with the Cockcroft-Gault formula.
5. Seropositivity for HBs Ag, HCV Ab, HIV 1 or HIV 2 Ab.
6. Any history of alcohol or drug abuse, or addiction within the last 2 years prior to enrollment.
7. Positive drug screening (opiates, cannabinoids, cocaine, methadone, amphetamines, barbiturates, ecstasy).
8. Positive alcohol or cotinine test.
9. Donation of blood, plasma or platelets within 3 months prior to the Screening visit or donation planned during the 3 months following the study.
10. Regular consumption of grapefruit juice or beverages containing xanthine bases (coffee, tea, cola: more than 5 cups or glasses a day).
11. Current smokers or smoking history < 6 months.
12. Current participation or participation within 3 months prior to the Screening visit, in another investigational drug or device study, or previous enrolment in the present study.
13. Chronic use of any drugs (prescription or over the counter [OTC]) within 4 weeks prior to enrollment (single use of medication such as paracetamol for headache is allowed, except during the week before enrollment).
14. Use of antioxidant vitamin supplements within 1 week prior to enrollment.
15. Use of mouthwash or toothpaste containing chlorhexidine within 1 week prior to randomization (applicable only for study Part 1).
16. In custody due to an administrative or a legal decision, or under tutelage, or being admitted to a sanitary or social institution.
17. Any direct or indirect involvement with the study conduct or staff at site or any family link with study site staff.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Part 1 : PK profile in plasma, saliva and urine : determination of nitrate levels. | from Day 1 morning to Day 7 morning .
Part 2 : PK profile in plasma : assess the Gamma-Hydroxybutyric acid (GHB) levels | Day 1 to Day 4

SECONDARY OUTCOMES:
Part 1: PK profile in saliva : determination of nitrite levels | from Day 1 morning to Day 7 morning .
Part 2 : PK profile in plasma : determination of nitrate levels | Day 1 to Day 4
Part 1 : PK profile in plasma : determination of Gamma-Hydroxybutyric acid (GHB) levels | from Day 1 morning to Day 7 morning
Part 1 : PK profile in plasma : determination of 1,4-butanediol mononitrate (BDMN) levels | from Day 1 morning to Day 7 morning
Part 1 : PK profile in plasma : determination of naproxcinod levels | from Day 1 morning to Day 7 morning
Part 1 : PK profile in plasma : determination of naproxen levels | from Day 1 morning to Day 7 morning
Part 1 : PK profile in urine : determination of nitrosoproline levels | from Day 1 morning to Day 7 morning
Part 1 : assess the general safety and tolerability | from Day 1 morning to Day 7 morning
Part 2 : PK profile in plasma: determination of BDMN levels | Day 1 to Day 4
Part 2 : PK profile in plasma : determination of naproxcinod levels | Day 1 to Day 4
Part 2 : PK profile in plasma: determination of naproxen levels | Day 1 to Day 4
Part 2 : assess the general safety and tolerability | Day 1 to Day 4

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rusca, MD FMH, Principal Investigator — Cross Research S.A. Phase I Unit

REFERENCES:
- See also: Nicox web-site — http://www.nicox.com